CLINICAL TRIAL: NCT06999382
Title: Contextually Responsive Implementation of Place Activation Interventions for Promoting Physical Activity in Marginalized Urban Peripheries in Mexico
Brief Title: Place Activation in Urban Peripheries: the 'Comunidades y Espacios Activos" Project (CEA)
Acronym: CEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); The University of Texas Health Science Center, Houston (Other); Washington University School of Medicine (Other); Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UTexasAustin-STUDY00005076; R01MD019155 (NIH)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Uptake of Systematic Review Evidence
Keywords: dissemination and implementation; place-activation; urban health; built environment; physical activity; contextual adaptations
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active 'Dissemination and Implementation' Place-Activation Intervention (Experimental): Intervention conditions include capacity-building activities for participants (who are defined as "implementation partners" - i.e., local stakeholders/decision makers and community leaders in the intervention neighborhoods), as well as evidence-based intervention implementation support for 1-year, which are hypothesized to improve adoption, reach, and fidelity of place-activation evidence-based interventions in urban settings. Activities include workshops, facilitation of coalition building activities, newsletters, targeted messaging, and access to a knowledge broker.
  Interventions: Behavioral: Active Dissemination and Implementation
- Comparison (Active Comparator): Implementation Partners in neighborhoods randomized to the active comparator arm will receive a booklet denominated a "menu of evidence-based interventions for place-activation to promote physical activity in urban settings", summarizing evidence-based approaches known to work to activate recently renovated or added public open spaces. They will also receive a pamphlet with information on the importance of healthy lifestyle promotion.
  Interventions: Behavioral: Passive Dissemination

INTERVENTIONS:
Behavioral: Active Dissemination and Implementation — This intervention is designed to accelerate the uptake of evidence-based interventions that help maximize the impact of the addition or renovation of public open spaces on their utilization for active recreation among community members, ultimately effective physical activity levels in communities. The intervention targets implementation partners: local stakeholders/decision makers and community leaders, to increase their awareness of these evidence-based approaches for place-activation, and their willingness to adopt and implement them in their neighborhood settings. Intervention components include capacity building workshops, newsletters, targeted messaging and access to a knowledge broker and implementation support for 1-year.
  Arms: Active 'Dissemination and Implementation' Place-Activation Intervention
Behavioral: Passive Dissemination — Delivery of booklet with menu of evidence-based interventions for place-activation; and of pamphlet summarizing importance of healthy lifestyle promotion.
  Arms: Comparison

SUMMARY:
This study will use a Hybrid III Cluster-Randomized Controlled Trial to test an 'active dissemination and implementation' intervention in peripheral urban neighborhoods, designed to accelerate the uptake of evidence-based place-based activations that are known to be effective in increasing physical activity among local residents. The study will use a parallel design with eligible neighborhoods randomized to one of two arms: the (1) "Active Dissemination and Implementation" intervention arm (n=15 neighborhoods); and (2) the comparison arm (n=15 neighborhoods). Participants will be "implementation partners" in each of the participating neighborhoods (n=510 total participants, n=17 per neighborhood), comprised of a mix of local government representatives, representatives of non-governmental organizations working in the area, and community leaders. Intervention components to be delivered to implementation partners of neighborhoods randomized to the "Active Dissemination and Implementation" Intervention Arm include participation in 2 workshops, facilitation of coalition building activities, newsletters, targeted messaging, and access to a knowledge broker, and implementation support for 1 year (12 months).

DETAILED DESCRIPTION:
A group-randomized hybrid III trial (Aim 2) testing the effectiveness of a 1-year 'active dissemination and implementation' intervention in increasing the reach, adoption, and implementation fidelity (primary outcomes); and the real-world effectiveness (secondary outcome) of contextually relevant place-activation evidence-based interventions. 30 urban peripheral neighborhoods with recently completed open public space improvements will be selected and randomized within pairs to the intervention vs. comparison condition (15 in each arm). Participants (n=510 total, n=17 per neighborhood) will be community leaders and local-level stakeholders with authority over or engagement with the public open space being assessed. Intervention conditions include capacity-building activities for participants, and intervention implementation support for 1-year, which are hypothesized to improve adoption, reach, and implementation fidelity of place-activation evidence-based interventions.

ELIGIBILITY:
Inclusion Criteria for Implementation Partners (main sample for primary Outcomes):

* Adults 18 years of age or older
* Stakeholders (government or nongovernmental organization representatives in sectors such as health, education, air quality, economic development, urban planning, transportation, parks and recreation, public safety, etc.) or community leaders of peripheral urban neighborhoods of study cities (10 possible cities in Mexico: Colima, Merida, Monterrey, Toluca, Mexico City, Guadalajara, Tijuana, Leon, Cuernavaca, Tapachula).

Exclusion Criteria for Implementation Partners (main sample of primary outcomes):

* Not meeting any of the inclusion criteria.

Inclusion Criteria for Intercept Survey Participants (for secondary outcomes):

* 18 years or older
* Located within the confines of the public open space being assessed in a study neighborhood at time of direct observation assessments.

Exclusion Criteria for Intercept Survey Participants (for secondary outcomes):

* Not meeting any of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Reach | Measured at baseline, 6-months (interim effects), 12-months (post-intervention), 24-months (maintenance)
  Operationalized as awareness of evidence-based interventions, and measured with surveys utilizing 5-Point Likert scale questions (Range: 1-5, where 5 is highest awareness).
Adoption (self-reported by implementation partners) | Measured at baseline, 6-months (interim effects), 12-months (post-intervention), 24-months (maintenance)
  Operationalized as the confirmed adoption of evidence-based interventions (binary variable: yes or no for each evidence-based intervention that could be adopted). Confirmation of adoption is assessed via surveys to implementation partners, who respond to questions about whether the neighborhood they operate at has begun utilizing each of the specific evidence-based interventions or not.
Implementation (self-reported) | Measured at baseline, 6-months (interim effects), 12-months (post-intervention), 24-months (maintenance)
  Operationalized as implementation fidelity, as reported by the implementation partner participants - i.e., to what extent is each of the evidence-based interventions that were adopted in a given neighborhood been implemented with close fidelity to the research-based intervention with proven effectiveness per the scientific literature. Implementation fidelity is measured with self-reported checklists.

SECONDARY OUTCOMES:
Adoption (group-level) | Measured at baseline, 6-months (interim effects), 12-months (post-intervention), 24-months (maintenance)
  Operationalized as confirmed adoption of evidence-based interventions at the neighborhood level. Assessed via policy document audits that my indicate a new program in place in the area or budget allocation for a given program; as well as by direct observation of public open spaces to confirm that a given intervention is taking place; and through intercept surveys to fully identifiable public open space users that report if to their knowledge any evidence-based intervention is ongoing in their neighborhood (analyzed at the group level for the given public open space where data were collected at each time point).
Implementation (group-level) | Measured at baseline, 6-months (interim effects), 12-months (post-intervention), 24-months (maintenance)
  Operationalized as the extent to which evidence-based interventions that have been adopted in a given neighborhood are taking place with close fidelity to the interventions that were developed and tested in research settings as reported by peer-reviewed literature. Measured via direct observation of public open spaces in participating neighborhoods, through direct observation checklists.
Real world effectiveness (physical activity) | Measured at baseline, 6-months (interim effects), 12-months (post-intervention), 24-months (maintenance)
  Measured by direct observation of public open spaces in participating neighborhoods, through the System for Observing Play and Recreation in Communities (SOPARC), a valid and reliable method utilizing spatial and momentary sampling assessments, measuring the number of total and physically active users of public open spaces. These data are then used to estimate group-based MET-minutes at a given point in space and time.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Salvo, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- Instituto Nacional de Salud Publica, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Longitudinal prospective data on a cohort of 510 community members and stakeholders, with measurements at baseline, and follow-ups at 6, 12, and months, will be collected using questionnaires. In addition, the project will provide longitudinal observation data collected annually in 30 public open spaces and cross-sectional panel data from up to 4,500 intercept surveys across the study duration (24 months).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available at the time of associated publication. The data submission and release timeframes specified by the funding agency and policies, as described on NIH's data sharing webpage, will be met. Study data deposited in the indicated repository or repositories will be available to the research community for a minimum of 7 years post-project end period or as long as administratively valuable per UT Austin data retention policies, plus any additional time required by the specific funding agency.
Access Criteria: Datasets will be findable and identifiable in ICPSR's database through a study digital object identifier (DOI) minted by ICPSR.